CLINICAL TRIAL: NCT00740311
Title: Comparative Clinical Study of the Prevention of the Reduction of Alveolar Crest by Alveoli Filling With an Injectable Calcium Phosphate After Extraction of Mandibular Molar or Pre Molar
Brief Title: Filling of Tooth Sockets With MBCP Gel TM Versus Technical Without Filling
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Other Study IDs: BRD06/9-O
Record Dates: First submitted 2008-08-21; First posted 2008-08-22 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-06

CONDITIONS: Alveolar Crest
Keywords: Prevention of the reduction of the alveolar crest

ARMS (2):
- Filling (Experimental): alveoli filling with an injectable calcium phosphate after extraction of mandibular molar or pre molar
  Interventions: Device: MBCP gel TM
- Without filling (No Intervention)

INTERVENTIONS:
Device: MBCP gel TM — alveoli filling with an injectable calcium phosphate after extraction of mandibular molar or pre molar
  Arms: Filling

SUMMARY:
After a dental extraction, the osseous alveoli fill naturally of a blood clot which is transformed some month later into osseous tissues. Even if the alveolar walls remain intact at the end of the intervention, the healing always comes along with a physiological reduction at the level of the site. The reduction of the alveolar crests is a continuous, cumulative and inexorable phenomenon This reduction entails in the long term aesthetic and functional damages which complicate the prosthetic rehabilitation of the dental articulate. That the prosthetic rehabilitation is removable or fixed, implanto-carried or not, it is made more difficult and less comfortable for the patient. In oral surgery, certain pathologies require for their treatment the use of materials of filling generating an activity of reduction / osseous replacement ending in the formation of a physiological calcified neo-tissue. Numerous products of osseous replacement were already used to realize alveolar fillings to avoid this inevitable and strongly harmful osseous loss.The purpose of the present study is to quantify the physiological osseous loss due to the dental extraction with or without filling by a randomized study and with calibrated criteria of evaluation. The current standard of care is no filling (healing from the blood clot) and we know the consecutive osseous loss during the aging. The technique by filling with an osseous substitute is more and more used in Europe and in Asia because of the decrease of the osseous loss. At first, these substitutes were constituted by bone grafts (autografts, allografts, xenografts) that tend to be replaced by synthetic materials. To realize these fillings according to countries, various materials are used (bovine bone, coral, bio glasses, phosphates of calcium). The most used synthetic materials are calcium ortho phosphates, the composition of which is close to mineral phases of calcified tissues. Ceramic of phosphate of calcium and more particularly the Biphasic Phosphate Calcium (BCP) was already used in numerous clinical applications.We chose as this study MBCP gel ™, same product beforehand used in 2 clinical studies for which the Nantes University Hospital was the sponsor.The perspectives of this study are to be able to propose the systematization of the alveolar filling to be able to decrease the osseous reduction after an extraction and to be able to propose more functional prosthetic rehabilitation (improvement of the masticatory power), more aesthetic and comfortable. When we know the effect of the under nutrition due to masticator difficulties notably at the aged persons, we measure all the importance of this major problem of Public health.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged from 18 to 75 years, in good general health
* Affiliated to a national insurance scheme or a beneficiary such a regime, having had a preliminary medical examination
* Without clinically significant buccal pathology or significant buccal concomitant treatment
* Presenting at least a mandibular embedded premolar or molar not conservable (maximum 3 molars or premolars not conservable, and no akin tooth),

Exclusion Criteria:

* Emergency extraction, or extraction that should not entail an osseous resorption other than a physiological one
* Lacteal tooth
* Trophic lesion
* Acute or chronic osteomyelitis, cellulitis, dry or infectious sachet non treated, granuloma or cyst not treated
* Filling revised surgical site with non resorbable biomaterial waste
* Filling necrotic surgical site
* Opening of brains
* Past or planned cervicofacial irradiation
* Known addiction to tobacco and alcohol
* Patient that hasn't a sufficient oral hygiene and which could not be better
* Allergy to Spiramycine, Metronidazole, Hydroxyzine, Paracetamol, Dextropropoxyphene, Chlorhexidine, or components of the local anesthesia
* Cancer, non equilibrate diabetes, tuberculosis, evolutionary or non equilibrate infectious or inflammatory disease
* Degenerative osseous pathology
* Distance infection risk
* Immunodeficiency
* Corticoids or other treatment with an effect on phosphocalcic metabolism
* Expectant mothers, parturients and the mothers who nurse (efficient contraception is mandatory).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-11; Primary Completion 2010-11 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is to compare the reduction of the alveolar crest with or without alveoli filling, verifying if the height of the filled alveolar crests is higher after 3 or 6 month compared to the height of the unfilled alveolar crests.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier universitaire, Nantes, France